CLINICAL TRIAL: NCT00507728
Title: Pharmacogenetics, Emotional Reactivity and Smoking
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-1024; 1R01DA017073 (NIH); NCI-2012-02108 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Results first posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Tobacco Use Disorder; Smoking Cessation
Keywords: Pharmacogenetics; Emotional Reactivity; Smoking Cessation Counseling; Smoking; Bupropion; Wellbutrin; Wellbutrin SR; Zyban; Varenicline; Chantix; Placebo
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Smoking | interventions — Bupropion; Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bupropion (Experimental): Bupropion starting dose 150 mg by mouth daily (150 mg every morning for three days; 150 mg twice a day thereafter).
  Interventions: Drug: Bupropion; Behavioral: Smoking Cessation Counseling
- Varenicline (Experimental): Varenicline starting dose 0.5 mg by mouth daily (0.5 mg every morning for days 1 - 3, then 0.5 mg twice a day for days 4 - 7, then 1 mg twice a day thereafter).
  Interventions: Drug: Varenicline; Behavioral: Smoking Cessation Counseling
- Placebo (Placebo Comparator): Placebo by mouth for 12 weeks.
  Interventions: Drug: Placebo; Behavioral: Smoking Cessation Counseling

INTERVENTIONS:
Drug: Bupropion — Starting dose 150 mg by mouth daily (150 mg every morning for three days; 150 mg twice a day thereafter)
  Other Names: Wellbutrin; Wellbutrin SR; Zyban
  Arms: Bupropion
Drug: Varenicline — Starting dose 0.5 mg by mouth daily (0.5 mg every morning for days 1 - 3, then 0.5 mg twice a day for days 4 - 7, then 1 mg twice a day thereafter)
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — Placebo by mouth for 12 weeks.
  Arms: Placebo
Behavioral: Smoking Cessation Counseling — Counseling over 8 months and telephone support calls.

SUMMARY:
The goals of this placebo-controlled randomized clinical trial were to evaluate the differences in emotional reactivity (peak startle response to affective stimuli) during a cessation attempt among smokers treated with bupropion, varenicline, or placebo, and to determine if these differences were moderated by genotype.

DETAILED DESCRIPTION:
Bupropion and Varenicline are smoking cessation aids that may help people to quit smoking.

During the orientation visit, the study will be explained to you and you will be given an opportunity to ask, and have answered, any questions you may have. You will also be asked to give a buccal (cheek cell) sample for genetic analysis. This session will last about 1.5 hours.

During the screening visit, you will be asked questions about your health, medication use, smoking history, and tobacco use. You will be asked about any current or past feelings of depression. Also, a small blood sample will be drawn (about 2 tablespoons) from your upper arm for a liver and kidney function test and a saliva sample will be collected to measure whether you are smoking. Women who are able to have children must have a negative urine pregnancy test. This session will last about 2.5 hours.

If you are eligible to take part in the study, you will be randomly assigned (as in the toss of a coin) to one of three treatment groups. Participants in the first group will receive Bupropion. Participants in the second group will receive Varenicline. Participants in the third group will receive a placebo. A placebo is a substance that looks like the study drug but which has no active ingredients. You will have an equal chance of being assigned to the Bupropion, Varenicline, or placebo treatment group. Neither you nor your counselor will know to which group you were assigned.

All participants will take study pills (either Bupropion, Varenicline, or placebo) by mouth for 12 weeks. The dose of study medication may or may not change during the study. You will be responsible for returning any unused, used, or partly used study medication bottles to a study staff member.

All participants will receive smoking cessation counseling to help them quit smoking, in the form of both in-person and telephone counseling sessions. Some of the counseling sessions may be videotaped or audio-taped. The videotapes will be used to help the investigators make sure that the counselors are following the correct procedures and will be erased within one year following your completion of the study. No one but the study investigators or those delegated by the study investigators will be allowed to view the tapes and the identity of the participants will be kept strictly confidential. Staff that may be given permission to view the tapes include project staff, consultants that review and rate how well the study counselors follow guidelines, and/or consultants that review how well the assessments are given.

You will need to come to the Behavioral Science Research Clinic at M. D. Anderson for 9 clinic visits over an 8-month period. You will receive 5 telephone calls from the study staff (while in treatment and during follow-up) to check on your progress in quitting smoking.

You will complete your first lab evaluation session (baseline) before any treatment begins (while you are still smoking). Immediately after the baseline lab session (on the same day), you will begin to receive counseling to quit smoking. You will begin taking one of the 3 study medications (Bupropion, Varenicline, or placebo) the next morning.

There will be 3 lab sessions, during which you will be asked to complete questionnaires about your mood and feelings (about 30 minutes total). Also, you will give a breath sample by blowing air into a small tube. This sample shows how much you have smoked. In each session you will be asked to watch slides and listen to a series of tones through earphones. The slides will include pictures of people, nature scenes, and artwork. Slides showing victims of car crashes, medical procedures, and nude people will also be shown. You will be shown examples of these slides before beginning the procedure and given the opportunity to withdraw from the study. During the lab sessions, your heart rate, brain electrical activity (EEG), skin sweating, and muscle tension will be monitored. To do this, small sensors will be placed on the fingers, arms, scalp and face. You should not drink more than 2 cups of coffee or other caffeine drinks at least 2.5 hours before each session.

During the first counseling visit, you will set a quit date for stopping smoking about 2 weeks after starting your study medication. You are asked not to quit smoking before the set quit date. After your quit date, you are asked to stay smoke free. You are asked to attend all your sessions whether you are smoking or not. All participants will receive smoking cessation counseling in the form of both in-person and telephone counseling sessions. The purpose of these visits will be to prepare you for quitting and to check the effects of the study medication on your attempt to stop smoking.

At each of your clinic visits, your blood pressure will be taken and you will be asked to blow air through a carbon monoxide (CO) measuring device. CO is a gas that is found in higher levels among cigarette smokers. At several visits you will be asked to provide a saliva sample to check for cotinine, a chemical produced by the breakdown of nicotine during smoking. You will be asked to give a saliva sample in a collection tube. Like the CO test, this test will help researchers measure how much you are smoking.

At your visits you will be asked questions about your smoking behavior. You will also be asked questions about your health and medical condition, and about any medications you are taking. You will be asked to complete a daily diary on cigarette smoking and drug dosing.

You will also be asked to mail saliva samples back to the clinic at least two times after stopping the medication. This will allow researchers to check on your smoking status.

Your total participation in this study will last about 8 months. This will include a 3-month and 6-month follow-up visit after your scheduled quit date. If the study staff is not able to reach you by phone, mail, or the information provided by your contacts, they may try to locate you through telephone directory assistance (411) or internet search sources (for example, Google or Yahoo!), which use information from the public domain (meaning everyone has access to it). If the study staff is still unable to find you, they may use a locator service such as Transunion or the National Change of Address (NCOA) database maintained by the United States Postal Service, as a last resort. Transunion uses magazine subscriptions and credit applications to find new addresses, and the NCOA uses the Change of Address cards filed with the post office when a person moves and requests their mail be forwarded to a new address. If the study staff has to use either of these services, they would only disclose your name and last known address.

At the end of the study, you will be able to ask additional questions about the results of the study and about procedures you have experienced during the study. Additionally, you will be able to sign up to receive a copy of the paper that will be written at the completion of the study.

This is an investigational study. Up to 375 smokers will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years old
2. Smoking: >/= 5 cigarettes per day within the 2 months preceding the screening visit and expired CO greater than or equal to 6 ppm.
3. Able to follow verbal and written instructions in English and complete all aspects of the study
4. Have an address and home telephone number where they may be reached
5. Provide informed consent and agree to all assessments and study procedures
6. Be the only participant in their household

Exclusion Criteria:

1. Within the month immediately preceding the screening visit; use of any form of tobacco product other than cigarettes on 3 or more days within a week only if the individual refuses to refrain from non-cigarette tobacco use during the course of this study
2. Within the month immediately preceding the screening visit; use of marijuana in any form on 3 or more days within a week
3. Within the two weeks immediately preceding the screening visit, involvement on more than 3 days in any formal smoking cessation activities
4. Current visual or auditory problems that in the opinion of the investigator would interfere with the completion of study assessments
5. Treatment on a continuous basis within 2 weeks before the screening visit: any contraindicated medication for Varenicline or Bupropion.
6. Uncontrolled hypertension or other major contraindications for Bupropion or Varenicline.
7. Severe renal impairment (CR Clearance <30 ml/min/1.73 m2).
8. Laboratory evaluations outside normal limits and of potential clinical significance in the opinion of the investigator
9. Meet current criteria for psychiatric disorders or substance abuse as assessed by the MINI for items A, B, D, I, J, K, L, M and N, including a past manic or hypomanic episode as well as a lifetime psychotic disorder.
10. Subject rated as moderate to high on suicidality as assessed by the MINI.
11. Psychiatric hospitalization within 1 year of screening date.
12. A positive urine pregnancy test during the screening period. Women who are two years post menopausal, one year post-tubal ligation, or who have had a partial or full hysterectomy will not be subject to a urine pregnancy test.
13. Pregnant, breast-feeding, or of childbearing potential who is not protected by a medically acceptable, effective method of birth control while enrolled in the study
14. Use of Varenicline or Bupropion within two weeks before the screening visit.
15. History of hypersensitivity or allergic reaction to Varenicline, tricyclic antidepressant, Bupropion (Wellbutrin, Zyban) or similar chemical classes or any component of these formulations.
16. Subject considered by the investigator as unsuitable candidate for receipt of an investigational drug, or unstable to be followed up throughout the entire duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2005-12-08 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cinciripini, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Cui Y, Robinson JD, Versace F, Lam CY, Minnix JA, Karam-Hage M, Dani JA, Kosten TR, Wetter DW, Brown VL, Cinciripini PM. Differential cigarette-related startle cue reactivity among light, moderate, and heavy smokers. Addict Behav. 2012 Aug;37(8):885-9. doi: 10.1016/j.addbeh.2012.02.003. Epub 2012 Feb 15. PMID 22571920
- [Background] Cui Y, Versace F, Engelmann JM, Minnix JA, Robinson JD, Lam CY, Karam-Hage M, Brown VL, Wetter DW, Dani JA, Kosten TR, Cinciripini PM. Alpha oscillations in response to affective and cigarette-related stimuli in smokers. Nicotine Tob Res. 2013 May;15(5):917-24. doi: 10.1093/ntr/nts209. Epub 2012 Oct 11. PMID 23060019
- [Background] Cui Y, Robinson JD, Engelmann JM, Lam CY, Minnix JA, Karam-Hage M, Wetter DW, Dani JA, Kosten TR, Cinciripini PM. Reinforcement sensitivity underlying treatment-seeking smokers' affect, smoking reinforcement motives, and affective responses. Psychol Addict Behav. 2015 Jun;29(2):300-311. doi: 10.1037/adb0000050. Epub 2015 Jan 26. PMID 25621416
- [Background] Cui Y, Engelmann JM, Xian J, Minnix JA, Lam CY, Karam-Hage M, Cinciripini PM, Robinson JD. Pharmacological intervention and abstinence in smokers undergoing cessation treatment: A psychophysiological study. Int J Psychophysiol. 2018 Jan;123:25-34. doi: 10.1016/j.ijpsycho.2017.12.001. Epub 2017 Dec 6. PMID 29223599
- [Background] Minnix JA, Versace F, Robinson JD, Lam CY, Engelmann JM, Cui Y, Brown VL, Cinciripini PM. The late positive potential (LPP) in response to varying types of emotional and cigarette stimuli in smokers: a content comparison. Int J Psychophysiol. 2013 Jul;89(1):18-25. doi: 10.1016/j.ijpsycho.2013.04.019. Epub 2013 May 2. PMID 23643564
- [Background] Robinson JD, Versace F, Lam CY, Minnix JA, Engelmann JM, Cui Y, Karam-Hage M, Shete SS, Tomlinson GE, Chen TT, Wetter DW, Green CE, Cinciripini PM. The CHRNA3 rs578776 Variant is Associated with an Intrinsic Reward Sensitivity Deficit in Smokers. Front Psychiatry. 2013 Sep 23;4:114. doi: 10.3389/fpsyt.2013.00114. eCollection 2013. PMID 24065931
- [Background] Versace F, Minnix JA, Robinson JD, Lam CY, Brown VL, Cinciripini PM. Brain reactivity to emotional, neutral and cigarette-related stimuli in smokers. Addict Biol. 2011 Apr;16(2):296-307. doi: 10.1111/j.1369-1600.2010.00273.x. Epub 2010 Dec 23. PMID 21182573
- [Background] Versace F, Lam CY, Engelmann JM, Robinson JD, Minnix JA, Brown VL, Cinciripini PM. Beyond cue reactivity: blunted brain responses to pleasant stimuli predict long-term smoking abstinence. Addict Biol. 2012 Nov;17(6):991-1000. doi: 10.1111/j.1369-1600.2011.00372.x. Epub 2011 Oct 4. PMID 21967530
- [Background] Versace F, Engelmann JM, Robinson JD, Jackson EF, Green CE, Lam CY, Minnix JA, Karam-Hage MA, Brown VL, Wetter DW, Cinciripini PM. Prequit fMRI responses to pleasant cues and cigarette-related cues predict smoking cessation outcome. Nicotine Tob Res. 2014 Jun;16(6):697-708. doi: 10.1093/ntr/ntt214. Epub 2013 Dec 27. PMID 24376278
- [Background] Meyer MJ, Coull BA, Versace F, Cinciripini P, Morris JS. Bayesian function-on-function regression for multilevel functional data. Biometrics. 2015 Sep;71(3):563-74. doi: 10.1111/biom.12299. Epub 2015 Mar 18. PMID 25787146
- [Background] Zhu H, Versace F, Cinciripini PM, Rausch P, Morris JS. Robust and Gaussian spatial functional regression models for analysis of event-related potentials. Neuroimage. 2018 Nov 1;181:501-512. doi: 10.1016/j.neuroimage.2018.07.006. Epub 2018 Jul 6. PMID 30057352
- [Background] Cinciripini PM, Green CE, Robinson JD, Karam-Hage M, Engelmann JM, Minnix JA, Wetter DW, Versace F. Benefits of varenicline vs. bupropion for smoking cessation: a Bayesian analysis of the interaction of reward sensitivity and treatment. Psychopharmacology (Berl). 2017 Jun;234(11):1769-1779. doi: 10.1007/s00213-017-4580-2. Epub 2017 Mar 8. PMID 28275830
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Cinciripini PM, Robinson JD, Karam-Hage M, Minnix JA, Lam C, Versace F, Brown VL, Engelmann JM, Wetter DW. Effects of varenicline and bupropion sustained-release use plus intensive smoking cessation counseling on prolonged abstinence from smoking and on depression, negative affect, and other symptoms of nicotine withdrawal. JAMA Psychiatry. 2013 May;70(5):522-33. doi: 10.1001/jamapsychiatry.2013.678. PMID 23536105
- [Derived] Versace F, Engelmann JM, Jackson EF, Costa VD, Robinson JD, Lam CY, Minnix JA, Brown VL, Wetter DW, Cinciripini PM. Do brain responses to emotional images and cigarette cues differ? An fMRI study in smokers. Eur J Neurosci. 2011 Dec;34(12):2054-63. doi: 10.1111/j.1460-9568.2011.07915.x. Epub 2011 Nov 20. PMID 22097928
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 254 subjects were randomized (varenicline: 75; bupropion: 89; placebo: 90 between December 2005 through October 2010. All subjects were residing in the Greater Houston Area and the study was completed at UT MD Anderson Cancer Center.
Pre-assignment Details: 646 participants signed consent, 392 were screen failures
Period: Randomization to Month 3
Arm/Group | Varenicline | Bupropion | Placebo
Started | 75 | 89 | 90
Completed | 60 | 75 | 70
Not Completed | 15 | 14 | 20
Not completed — Lost to Follow-up | 15 | 14 | 20
Period: From 3 Months to 6 Months
Arm/Group | Varenicline | Bupropion | Placebo
Started | 60 | 75 | 70
Completed | 54 | 65 | 61
Not Completed | 6 | 10 | 9
Not completed — Lost to Follow-up | 6 | 10 | 9

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all treated participants, i.e. Intention to Treat.
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Bupropion | Placebo | Total
Number analyzed (Participants) | 75 | 89 | 90 | 254
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.5 (10.8) | 44.5 (9.3) | 45.7 (10.9) | 44.6 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 34 | 34 | 98
  Male | 45 | 55 | 56 | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 7 | 24
  Not Hispanic or Latino | 63 | 82 | 80 | 225
  Unknown or Not Reported | 1 | 1 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Asian | 3 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 18 | 23 | 22 | 63
  White | 39 | 57 | 60 | 156
  More than one race | 10 | 4 | 6 | 20
  Unknown or Not Reported | 2 | 3 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 75 | 89 | 90 | 254
Demographic and individual-level characteristics Wisconsin Smoking Withdrawal Scale (WSWS) [Mean (Standard Deviation); unit: Score on a scale] — The Wisconsin Withdrawal Scale (WSWS) contains 7 factors: Anger, Anxiety, Sadness, Concentration, Craving, Sleep, and Hunger. WSWS consists of 28 items that are scored on a 5-point Likert type scale (0 = strongly disagree, 4 = strongly agree). Higher values, of all scales, represent worse outcomes
  Score on a scale
    WSWS Anger Subscale | 3.8 (2.6) | 4.2 (2.7) | 4.2 (7.9) | 4.1 (2.6)
    WSWS Anxiety Subscale | 7.3 (2.7) | 7.3 (3.2) | 7.9 (3.3) | 7.5 (3.1)
    WSWS Concentration Subscale | 3.7 (1.9) | 4 (2.2) | 3.9 (2.2) | 3.9 (2.1)
    WSWS Craving Subscale | 8.7 (3.1) | 9.4 (2.8) | 9.1 (2.6) | 9.1 (2.8)
    WSWS Hunger Subscale | 9.6 (3.7) | 9.8 (3.3) | 11.2 (3.7) | 10.2 (3.6)
    WSWS Sadness Subscale | 4.6 (2.5) | 4.2 (2.4) | 4.7 (2.5) | 4.5 (2.8)
    WSWS Sleep Subscale | 7.7 (4.3) | 9.3 (4.5) | 8.6 (4.4) | 8.6 (4.5)
Demographic and individual-level characteristics -Positive and Negative Affect Scales (PANAS) [Median (Standard Deviation); unit: Score on a scale] — The Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much). Scores can range from 10-50 for both the Positive and Negative Affect with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect
  Score on a scale
    PANAS Positive Affect | 35.8 (7.1) | 36.1 (5.7) | 35.8 (6.2) | 35.9 (6.3)
    PANAS Negative Affect | 14.8 (5.1) | 15.6 (6.9) | 16.4 (5.9) | 15.6 (5.3)
Demographic and individual-level characteristics - (CESD) [Mean (Standard Deviation); unit: Score on a scale] — Center of Epidemiologic Studies Depression Scale (CESD) a 20-item measure that asks caregivers to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
  Score on a scale | 6.7 (6.1) | 6.9 (6.1) | 8.1 (7.1) | 7.3 (6.5)
Demographic and individual-level characteristics -Modified Cigarette Evaluation Questionnaire (mCEQ) [Median (Standard Deviation); unit: scores on a scale] — Modified Cigarette Evaluation Questionnaire (mCEQ). mCEQ Smoking satisfaction: range (1-21); mCEQ Psychological Reward: range(1-35); mCEQ Aversion: range (1-14); mCEQ Enjoyment of Resp.Tract Sens: range (1-7); mCEQ Craving Reduction: range (1-7). For all scales of mCEQ higher scores indicate worse outcomes (greater intensity of smoking effect). Scores of mCEQ Smoking satisfaction, mCEQ psychological reward and mCEQ aversion were summed to create the subscales. mCEQ Enjoyment of Resp Tract Sens and mCEQ Craving Reduction were single items.
  scores on a scale
    mCEQ Smoking Satisfaction | 4.3 (1.1) | 3.9 (1.2) | 4.2 (1.2) | 4.2 (1.2)
    mCEQ Psychological Reward | 4.1 (4.9) | 3.7 (1.1) | 3.6 (1.3) | 3.8 (3.1)
    mCEQ Aversion | 1.6 (0.8) | 1.6 (0.7) | 1.5 (0.8) | 1.5 (0.8)
    mCEQ Enjoyment of Respiratory Tract Sensation | 2.9 (1.5) | 2.9 (1.4) | 2.9 (1.4) | 2.9 (1.5)
    mCEQ Craving Reduction | 5.1 (1.5) | 5.1 (1.4) | 4.9 (1.6) | 5 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Emotional Reactivity By Pharmacotherapy
Description: Emotional reactivity measured by the peak eye blink electromyography (EMG) of the orbicularis oculi (ORB) muscle responses to acoustic startle probe delivered during the presentation of emotionally valent stimuli (pleasant, unpleasant, neutral, and smoking-related pictures). A single value was estimated by averaging within the specific time interval.
Time Frame: Baseline to 1 month
Measure: Least Squares Mean (95% Confidence Interval); unit: microvolts
Arm/Group | Varenicline | Bupropion | Placebo
Number analyzed (Participants) | 78 | 89 | 90
microvolts
  Emotional Reactivity (ORB) to Cigarette Stimuli | 66.6 [62.3 to 71.1] | 64.7 [60.9 to 68.5] | 65.6 [61.5 to 69.7]
  Emotional Reactivity (ORB) to Negative Stimuli | 70.9 [66.4 to 75.4] | 73.1 [69.2 to 76.9] | 65.6 [61.5 to 69.7]
  Emotional Reactivity (ORB) to Positive Stimuli | 66.7 [62.5 to 70.9] | 65.4 [61.8 to 68.9] | 64.7 [60.8 to 68.6]
  Emotional Reactivity (ORB) to Neutral Stimuli | 59.6 [45.2 to 74.1] | 64.9 [52.7 to 77.2] | 72.5 [59.3 to 85.7]

2. Primary Outcome: Emotional Reactivity By Pharmacotherapy Moderated by DRD2 A1 Allele
Description: The emotional reactivity (ORB EMG) of smokers during cessation will be moderated by genotype. A single value was estimated by averaging within the specific time interval. During a quit attempt, smokers were evaluated on how they react to smoking related cues. An interaction term was then formed by the reactivity to smoking stimulus and genotype.
Time Frame: Baseline to 1 month
Population: 13 participants had missing data in DRD2 A1 and were not included in the analysis. 1 participant was from the Varenicline group, 7 from the Buproprion group and 5 from the placebo group.
Measure: Least Squares Mean (95% Confidence Interval); unit: microvolts
Groups:
- Varenicline w/o DRD2 A1 Allele: Subjects in the Varenicline group not carrying the DRD2 A1 allele
- Varenicline With DRD2 A1 Allele: Subjects in the Varenicline group carrying the DRD2 A1 allele
- Bupropion w/o DRD2 A1 Allele: Subjects in the Bupropion group not carrying the DRD2 A1 allele
- Bupropion With DRD2 A1 Allele; Placebo With DRD2 A1 Allele: Subjects in the Bupropion group carrying the DRD2 A1 allele
- Placebo w/o DRD2 A1 Allele: Subjects in the Placebo group not carrying the DRD2 A1 allele
Arm/Group | Varenicline w/o DRD2 A1 Allele | Varenicline With DRD2 A1 Allele | Bupropion w/o DRD2 A1 Allele | Bupropion With DRD2 A1 Allele | Placebo w/o DRD2 A1 Allele | Placebo With DRD2 A1 Allele
Number analyzed (Participants) | 48 | 26 | 37 | 45 | 41 | 44
microvolts
  Emotional Reactivity (ORB) to Cigarette Stimuli | 66.5 [61.1 to 71.9] | 69.9 [62.8 to 77.0] | 66.2 [60.4 to 72] | 66 [60.9 to 71.2] | 67.3 [61.5 to 73.1] | 68.1 [62.2 to 73.9]
  Emotional Reactivity (ORB) to Negative Stimuli | 70.5 [65 to 75.9] | 75.1 [67.9 to 82.2] | 78.6 [72.8 to 84.4] | 71.3 [66.2 to 76.5] | 74 [68.2 to 79.7] | 68.1 [62.2 to 73.9]
  Emotional Reactivity (ORB) to Positive Stimuli | 65.5 [60.4 to 70.6] | 72 [65.3 to 78.7] | 71.3 [65.8 to 76.7] | 63.3 [58.4 to 681.] | 68.5 [63.1 to 74] | 63.8 [58.3 to 69.4]
  Emotional Reactivity (ORB) to Neutral Stimuli | 55.3 [37.4 to 73.2] | 67.2 [43 to 91.5] | 73.9 [54.6 to 93.1] | 61.2 [44 to 78.3] | 79.7 [61 to 98.5] | 67.8 [48.3 to 87.2]

3. Secondary Outcome: Smoking Abstinence at 3 Months
Description: Values represent change in probability of abstinence for unit change in emotional reactivity. Abstinence data collected using a timeline follow-back (TLFB) procedure. Continuous Abstinence was defined as no smoking within the last 4 weeks of treatment. It is scored as 0 if the participant smoked during the specific interval, and 1 if the participant abstained from smoking.
Time Frame: Baseline to 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: probability
Arm/Group | Varenicline | Bupropion | Placebo
Number analyzed (Participants) | 75 | 89 | 90
probability
  Emotional Reactivity (ORB) to Cigarette Stimuli | -0.003 [-0.0777 to 0.072] | -0.01 [-0.084 to 0.065] | -0.008 [-0.096 to 0.081]
  Emotional Reactivity (ORB) to Negative Stimuli | -0.004 [-0.081 to 0.073] | -0.009 [-0.076 to 0.058] | -0.007 [-0.088 to 0.073]
  Emotional Reactivity (ORB) to Positive Stimuli | -0.003 [-0.081 to 0.076] | -0.01 [-0.084 to 0.064] | -0.007 [-0.092 to 0.079]
  Emotional Reactivity (ORB) to Neutral Stimuli | -0.004 [-0.085 to 0.076] | -0.008 [-0.084 to 0.068] | -0.007 [-0.088 to 0.075]

4. Secondary Outcome: Smoking Abstinence at 3 Months by DRD2 A1 Allele
Description: as for outcome 3
Time Frame: Baseline to 3 Month
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: probability
Arm/Group | Varenicline w/o DRD2 A1 Allele | Varenicline With DRD2 A1 Allele | Bupropion w/o DRD2 A1 Allele | Bupropion With DRD2 A1 Allele | Placebo w/o DRD2 A1 Allele | Placebo With DRD2 A1 Allele
Number analyzed (Participants) | 48 | 26 | 37 | 45 | 41 | 44
probability
  Emotional Reactivity (ORB) to Cigarette Stimuli | 0.001 [-0.002 to 0.004] | -0.004 [-0.008 to 0] | 0 [-0.003 to 0.003] | -0.003 [-0.006 to 0.001] | -0.001 [-0.003 to 0.001] | -0.004 [-0.008 to 0]
  Emotional Reactivity (ORB) to Negative Stimuli | 0.002 [-0.002 to 0.005] | -0.005 [-0.008 to -0.001] | 0 [-0.002 to 0.002] | -0.004 [-0.007 to 0.001] | -0.001 [-0.003 to 0.001] | -0.004 [-0.008 to 0]
  Emotional Reactivity (ORB) to Positive Stimuli | 0.001 [-0.002 to 0.005] | -0.005 [-0.009 to -0.001] | 0 [-0.003 to 0.002] | -0.003 [-0.006 to 0] | -0.001 [-0.003 to 0.001] | -0.004 [-0.007 to 0]
  Emotional Reactivity (ORB) to Neutral Stimuli | 0.001 [-0.002 to 0.005] | -0.005 [-0.009 to -0.001] | 0.001 [-0.002 to 0.003] | -0.002 [-0.005 to 0.001] | -0.001 [-0.003 to 0.001] | -0.003 [-0.007 to 0.001]

5. Secondary Outcome: Smoking Abstinence at 6 Months
Description: as for outcome 3
Time Frame: Abstinence at 6 Months ( the effects shown are the increase/decrease in probability of abstinence for 1 unit increase in the predictor)
Measure: Least Squares Mean (95% Confidence Interval); unit: probability
Arm/Group | Varenicline | Bupropion | Placebo
Number analyzed (Participants) | 75 | 89 | 90
probability
  Emotional Reactivity (ORB) to Cigaretee Stimuli | 0.007 [-0.067 to 0.082] | -0.002 [-0.073 to 0.069] | -0.006 [-0.091 to 0.079]
  Emotional Reactivity (ORB) to Negative Stimuli | 0.008 [-0.069 to 0.085] | -0.003 [-0.067 to 0.062] | -0.005 [-0.081 to 0.071]
  Emotional Reactivity (ORB) to Positive Stimuli | 0.01 [-0.065 to 0.086] | -0.003 [-0.075 to 0.068] | -0.005 [-0.087 to 0.078]
  Emotional Reactivity (ORB) to Neutral Stimuli | 0.008 [-0.071 to 0.087] | -0.001 [-0.078 to 0.076] | -0.005 [-0.052 to 0.041]

6. Secondary Outcome: Abstinence at 6 Months by DRD2 A1 Allele
Description: as for outcome 3
Time Frame: Baseline to 6 Month ( the effects shown are the increase/decrease in probability of abstinence for 1 unit increase in the predictor)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: probability
Arm/Group | Varenicline w/o DRD2 A1 Allele | Varenicline With DRD2 A1 Allele | Bupropion w/o DRD2 A1 Allele | Bupropion With DRD2 A1 Allele | Placebo w/o DRD2 A1 Allele | Placebo With DRD2 A1 Allele
Number analyzed (Participants) | 48 | 26 | 37 | 45 | 41 | 44
probability
  Emotional Reactivity (ORB) to Cigarette Stimuli | 0.003 [0 to 0.005] | -0.001 [-0.005 to 0.003] | 0.001 [-0.002 to 0.003] | -0.001 [-0.004 to 0.002] | 0 [-0.002 to 0.001] | -0.005 [-0.01 to 0]
  Emotional Reactivity (ORB) to Negative Stimuli | 0.003 [0.001 to 0.005] | -0.001 [-0.005 to 0.003] | 0.001 [-0.001 to 0.003] | -0.002 [-0.005 to 0.001] | 0 [-0.002 to 0.001] | -0.004 [-0.008 to 0]
  Emotional Reactivity (ORB) to Positive Stimuli | 0.003 [0.001 to 0.006] | 0 [-0.005 to 0.004] | 0 [-0.002 to 0.003] | -0.001 [-0.004 to 0.002] | 0 [-0.002 to 0.002] | -0.004 [-0.008 to 0]
  Emotional Reactivity (ORB) to Neutral Stimuli | 0.003 [0 to 0.005] | -0.001 [-0.005 to 0.003] | 0.001 [-0.002 to 0.004] | -0.001 [-0.004 to 0.002] | 0 [-0.002 to 0.001] | -0.004 [-0.009 to 0]

7. Secondary Outcome: Symptoms of Nicotine Withdrawal Using the Wisconsin Smoking Withdrawal Scale (WSWS)
Description: Symptoms of nicotine withdrawal measured using Wisconsin Smoking Withdrawal Scale (WSWS). The Wisconsin Withdrawal Scale (WSWS) contains 7 factors: Anger, Anxiety, Sadness, Concentration, Craving, Sleep, and Hunger. WSWS consists of 28 items that are scored on a 5-point Likert type scale (0 = strongly disagree, 4 = strongly agree). A single value was estimated by averaging within the specific time interval. Higher values represent worse outcome. The average value was estimated from Baseline to 8 months
Time Frame: Baseline to 8 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Varenicline w/o DRD2 A1 Allele | Varenicline With DRD2 A1 Allele | Bupropion w/o DRD2 A1 Allele | Bupropion With DRD2 A1 Allele | Placebo w/o DRD2 A1 Allele | Placebo With DRD2 A1 Allele
Number analyzed (Participants) | 48 | 26 | 37 | 45 | 41 | 44
score on a scale
  Anger | 4.394 [3.629 to 5.159] | 4.222 [3.152 to 5.291] | 4.28 [3.402 to 5.157] | 4.41 [3.59 to 5.23] | 5.584 [4.744 to 6.424] | 5.752 [4.884 to 6.621]
  Anxiety | 6.218 [5.384 to 7.052] | 5.873 [4.707 to 7.038] | 6.587 [5.63 to 7.543] | 6.587 [5.63 to 7.543] | 7.785 [6.87 to 8.7] | 7.915 [6.968 to 8.862]
  Concentration | 3.743 [3.117 to 4.369] | 3.407 [2.531 to 4.282] | 4.238 [3.521 to 4.956] | 3.935 [3.265 to 4.605] | 4.764 [4.077 to 5.451] | 4.951 [4.242 to 5.66]
  Craving | 6.646 [5.591 to 7.701] | 6.252 [4.777 to 7.726] | 6.814 [5.605 to 8.024] | 6.78 [5.651 to 7.91] | 9.024 [7.866 to 10.181] | 8.696 [7.499 to 9.893]
  Hunger | 11.016 [10.09 to 11.942] | 10.707 [9.413 to 12.001] | 9.79 [8.729 to 10.852] | 11.082 [10.09 to 12.074] | 11.207 [10.19 to 12.223] | 11.044 [9.994 to 12.095]
  Sadness | 4.246 [3.535 to 4.958] | 3.738 [2.744 to 4.732] | 4.005 [3.189 to 4.82] | 4.338 [3.577 to 5.1] | 5.293 [4.513 to 6.074] | 5.865 [5.057 to 6.673]
  Sleep | 7.721 [6.494 to 8.948] | 8.153 [6.438 to 9.868] | 9.672 [8.265 to 11.079] | 9.528 [8.214 to 10.843] | 9.078 [7.731 to 10.424] | 8.629 [7.236 to 10.023]

8. Secondary Outcome: Symptoms of Nicotine Withdrawal and Negative Affect Using Positive and Negative Affect Scale (PANAS)
Description: Symptoms of nicotine withdrawal and negative affect were measured using the Positive and Negative Affect Scale (PANAS). The Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much). Scores can range from 10-50 for both the Positive and Negative Affect with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect. The average value was estimated from Baseline to 8 months
Time Frame: Baseline to 8 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Varenicline w/o DRD2 A1 Allele | Varenicline With DRD2 A1 Allele | Bupropion w/o DRD2 A1 Allele | Bupropion With DRD2 A1 Allele | Placebo w/o DRD2 A1 Allele | Placebo With DRD2 A1 Allele
Number analyzed (Participants) | 48 | 26 | 37 | 45 | 41 | 44
score on a scale
  Positive Affect | 35.507 [33.494 to 37.521] | 37.315 [34.5 to 40.13] | 36.429 [34.122 to 38.735] | 35.281 [33.125 to 37.437] | 33.672 [31.463 to 35.882] | 33.984 [31.709 to 36.259]
  Negative Affect | 15.93 [14.404 to 17.455] | 14.98 [12.849 to 17.112] | 15.782 [14.032 to 17.532] | 16.385 [14.751 to 18.02] | 18.017 [16.343 to 19.691] | 18.902 [17.166 to 20.638]

9. Secondary Outcome: Symptoms of Depression Using the Center for Epidemiologic Studies Depression Scale (CES-D)
Description: Symptoms of nicotine withdrawal measured using Center for Epidemiologic Studies Depression Scale (CES-D). Center of Epidemiologic Studies Depression Scale (CESD) a 20-item measure that asks caregivers to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms. The average value was estimated from Baseline to 8 months
Time Frame: Baseline to 8 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Varenicline w/o DRD2 A1 Allele | Varenicline With DRD2 A1 Allele | Bupropion w/o DRD2 A1 Allele | Bupropion With DRD2 A1 Allele | Placebo w/o DRD2 A1 Allele | Placebo With DRD2 A1 Allele
Number analyzed (Participants) | 48 | 26 | 37 | 45 | 41 | 44
score on a scale | 8.084 [6.19 to 9.978] | 6.847 [4.2 to 9.494] | 7.588 [5.416 to 9.76] | 8.362 [6.333 to 10.39] | 8.65 [6.572 to 10.729] | 10.799 [8.647 to 12.951]

10. Secondary Outcome: Measures of Smoking Satisfaction and Psychological Reward Using the Modified Cigarette Evaluation Questionnaire (mCEQ) Subscales
Description: Modified Cigarette Evaluation Questionnaire (mCEQ). mCEQ Smoking satisfaction: range (1-21); mCEQ Psychological Reward: range(1-35); mCEQ Aversion: range (1-14); mCEQ Enjoyment of Resp.Tract Sens: range (1-7); mCEQ Craving Reduction: range (1-7). For all scales of mCEQ higher scores indicate worse outcomes (greater intensity of smoking effect). Scores of mCEQ Smoking satisfaction, mCEQ psychological reward and mCEQ aversion were summed to create the subscales. mCEQ Enjoyment of Resp Tract Sens and mCEQ Craving Reduction were single items.
Time Frame: Baseline to 8 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Varenicline w/o DRD2 A1 Allele | Varenicline With DRD2 A1 Allele | Bupropion w/o DRD2 A1 Allele | Bupropion With DRD2 A1 Allele | Placebo w/o DRD2 A1 Allele | Placebo With DRD2 A1 Allele
Number analyzed (Participants) | 48 | 26 | 37 | 45 | 41 | 44
score on a scale
  Smoking Satisfaction | 2.895 [1.912 to 3.879] | 2.591 [1.253 to 3.93] | 4.064 [2.94 to 5.187] | 3.369 [2.135 to 4.603] | 3.025 [2.087 to 3.963] | 3.515 [2.368 to 4.662]
  Psychological Reward | 2.819 [2.109 to 3.528] | 2.155 [1.181 to 3.13] | 2.519 [1.693 to 3.346] | 2.723 [1.812 to 3.634] | 3.575 [2.861 to 4.289] | 3.246 [2.399 to 4.093]
  Aversion | 1.612 [1.357 to 1.867] | 1.694 [1.342 to 2.045] | 1.988 [1.69 to 2.286] | 1.79 [1.461 to 2.119] | 1.808 [1.549 to 2.067] | 1.69 [1.384 to 1.996]
  Enjoyment of Respiratory Tract Sensation | 1.912 [0.146 to 3.678] | 1.703 [-0.692 to 4.099] | 4.096 [2.094 to 6.099] | 1.955 [-0.243 to 4.153] | 3.711 [2.048 to 5.375] | 2.783 [0.741 to 4.825]
  Craving Reduction | 4.531 [3.232 to 5.831] | 3.952 [2.2 to 5.705] | 4.564 [3.083 to 6.044] | 6.628 [5.017 to 8.238] | 4.486 [3.269 to 5.702] | 4.673 [3.176 to 6.17]

11. Secondary Outcome: Skin Conductance Response
Description: Skin conductance response (SCR) amplitude measured by placing an electrodermal response transducer on the fore and ring fingers of the participants non-dominant hand, and heart rate (HR) was collected by placing a photoelectric pulse plethysmogram transducer on the middle finger of the participants non-dominant hand, during the presentation of emotionally valent stimuli (positive, negative, neutral, and smoking-related pictures). A single value was estimated by averaging within the specific time interval.
Time Frame: Baseline to 1 month
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Microsiemens
Arm/Group | Varenicline w/o DRD2 A1 Allele | Varenicline With DRD2 A1 Allele | Bupropion w/o DRD2 A1 Allele | Bupropion With DRD2 A1 Allele | Placebo w/o DRD2 A1 Allele | Placebo With DRD2 A1 Allele
Number analyzed (Participants) | 48 | 26 | 37 | 45 | 41 | 44
Microsiemens
  Skin conductance to Cigarette Stimuli | 2.301 [1.619 to 2.982] | 2.016 [1.132 to 2.901] | 2.275 [1.512 to 3.037] | 1.797 [1.082 to 2.511] | 2.272 [1.54 to 3.005] | 2.443 [1.703 to 3.183]
  Skin conductance to Negative Stimuli | 2.295 [1.613 to 2.976] | 1.969 [1.084 to 2.855] | 2.31 [1.547 to 3.072] | 1.695 [0.999 to 2.391] | 2.355 [1.611 to 3.099] | 2.485 [1.756 to 3.215]
  Skin conductance to Positive Stimuli | 2.256 [1.58 to 2.931] | 1.984 [1.106 to 2.862] | 2.299 [1.542 to 3.055] | 1.7 [1.01 to 2.39] | 2.296 [1.569 to 3.023] | 2.565 [1.831 to 3.299]
  Skin conductance to Neutral Stimuli | 2.261 [1.578 to 2.944] | 2.017 [1.13 to 2.904] | 2.369 [1.602 to 3.136] | 1.699 [1.002 to 2.397] | 2.362 [1.616 to 3.107] | 2.559 [1.82 to 3.299]

12. Secondary Outcome: Heart Rate Response
Description: Heart Rate Response. A single value was estimated by averaging within the specific time interval. During a quit attempt, smokers were evaluated on how they react to smoking related cues. An interaction term was then formed by the reactivity to smoking stimulus and genotype.
Time Frame: Baseline to 1 month
Measure: Least Squares Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | Varenicline w/o DRD2 A1 Allele | Varenicline With DRD2 A1 Allele | Bupropion w/o DRD2 A1 Allele | Bupropion With DRD2 A1 Allele | Placebo w/o DRD2 A1 Allele | Placebo With DRD2 A1 Allele
Number analyzed (Participants) | 48 | 26 | 37 | 45 | 41 | 44
beats per minute
  Heart Rate response to Cigarette Stimuli | 69.731 [66.962 to 72.5] | 68.652 [65.068 to 72.236] | 71.427 [68.331 to 74.524] | 69.836 [66.974 to 72.699] | 65.966 [62.987 to 68.944] | 65.276 [62.266 to 68.286]
  Heart Rate response to Negative Stimuli | 69.562 [66.722 to 72.402] | 68.078 [64.403 to 71.753] | 71.077 [67.904 to 74.25] | 69.595 [66.699 to 72.492] | 65.768 [62.713 to 68.823] | 65.569 [62.523 to 68.615]
  Heart Rate response to Positive Stimuli | 69.151 [66.351 to 71.95] | 68.711 [65.087 to 72.334] | 71.518 [68.386 to 74.65] | 70.404 [67.546 to 73.262] | 65.787 [62.776 to 68.799] | 65.927 [62.929 to 68.926]
  Heart Rate response to Neutral Stimuli | 69.621 [66.798 to 72.444] | 68.969 [65.315 to 72.624] | 71.706 [68.546 to 74.865] | 70.234 [67.351 to 73.117] | 65.237 [62.2 to 68.273] | 66.04 [62.981 to 69.098]

ADVERSE EVENTS:
Time Frame: Baseline, up to 8 months
Arm/Group | Varenicline | Bupropion | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/89 | 0/90
Serious Adverse Events (participants affected / at risk) | 2/75 | 2/89 | 0/90
Other Adverse Events (participants affected / at risk) | 63/75 | 69/89 | 66/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=75) | Bupropion (N=89) | Placebo (N=90)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | 0
Increased Coughing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=75) | Bupropion (N=89) | Placebo (N=90)
ABSCESS (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
ACCIDENTAL INJURY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
APPETITE DECREASED (General disorders) | 3 | 4 | 3
APPETITE INCREASED (General disorders) | 8 | 7 | 5
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Abnormal Dreams (Psychiatric disorders) | 13 | 6 | 7
Allergic reaction (Immune system disorders) | 1 | 0 | 1
Allergy, Seasonal (Immune system disorders) | 1 | 2 | 1
Anxiety Symptoms (Psychiatric disorders) | 5 | 5 | 13
BLOOD IN STOOL (Gastrointestinal disorders) | 0 | 1 | 0
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
BRUISE (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Blurred vision (Eye disorders) | 1 | 4 | 2
Body odor (General disorders) | 1 | 0 | 0
Cerebrospinal fluid.. (Nervous system disorders) | 1 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 4 | 11
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Constipation (Gastrointestinal disorders) | 6 | 5 | 3
DIABETES MELLITUS (Endocrine disorders) | 0 | 0 | 1
Dehydration (General disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 6 | 7 | 10
Diarrhea (Gastrointestinal disorders) | 8 | 4 | 12
Disturbance in attention (Psychiatric disorders) | 7 | 7 | 12
Dizziness (General disorders) | 4 | 4 | 4
Drowsiness (Nervous system disorders) | 3 | 2 | 5
Dry mouth (General disorders) | 1 | 3 | 7
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 6 | 6 | 3
Edema (Musculoskeletal and connective tissue disorders) | 3 | 4 | 5
Elevated mood (Psychiatric disorders) | 0 | 0 | 1
Emotional liability (Psychiatric disorders) | 2 | 3 | 4
Eye irritation (Eye disorders) | 2 | 1 | 2
Fatigue (General disorders) | 4 | 5 | 9
Flatulence (Gastrointestinal disorders) | 2 | 4 | 1
Flushing (General disorders) | 1 | 0 | 2
Gastritis (Gastrointestinal disorders) | 6 | 5 | 4
Glucose intolerance (Endocrine disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 9 | 13 | 11
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Herniated Disc (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertension (Cardiac disorders) | 3 | 2 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Increased Coughing (Respiratory, thoracic and mediastinal disorders) | 9 | 7 | 4
Infection (General disorders) | 1 | 6 | 3
Influenza (General disorders) | 6 | 8 | 2
Insomnia (Nervous system disorders) | 16 | 26 | 13
Irritability (Psychiatric disorders) | 11 | 14 | 13
Kidney Stones (Renal and urinary disorders) | 0 | 1 | 0
Libido decreased (Reproductive system and breast disorders) | 0 | 1 | 0
Mucositis oral (General disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 9 | 12
Nausea (Gastrointestinal disorders) | 21 | 17 | 8
Neck pain (General disorders) | 1 | 2 | 1
PARESTHESIA (Nervous system disorders) | 1 | 0 | 1
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 2 | 6
Pelvic pain (General disorders) | 1 | 0 | 0
Reduced inhibition (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 5 | 5
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 17 | 26 | 23
SWEATING INCREASED (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Sensory disturbance (Nervous system disorders) | 1 | 0 | 2
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 11
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 9
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Surgical and medical (Surgical and medical procedures) | 1 | 0 | 0
TASTE PERVERSION (General disorders) | 4 | 3 | 6
TREMOR (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Tachycardia/Palpita.. (Cardiac disorders) | 1 | 3 | 0
Tinnitus (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Toothache (General disorders) | 3 | 7 | 3
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 3 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 2
Weight gain (General disorders) | 2 | 2 | 1
Weight loss (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2004-02-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT00507728/Prot_SAP_000.pdf